CLINICAL TRIAL: NCT06166264
Title: Effects of Progressive Resistance Training on Depression , Fatigue and Vasomotor Symptoms in Post Menopausal Women
Brief Title: Effects of Progressive Resistance Training Vasomotor Symptoms in Post Menopausal Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Principal Investigator, Adeela Arif, Senior Lecturer, Riphah International University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Saba Murtaza
Record Dates: First submitted 2023-12-04; First posted 2023-12-12 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Post Menopausal
Keywords: Depression; Fatigue; Vasomotor symptoms; Post-menopause
MeSH Terms: conditions — Depression; Fatigue | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Progressive resistance training (Experimental)
  Interventions: Other: Progressive resistance training
- Control group (Experimental)
  Interventions: Other: Control group

INTERVENTIONS:
Other: Progressive resistance training — It consists of patients who will receive both Resistance exercise training sessions and aerobic training 3 times per week for 8 weeks. Every session will be of 45 minutes. Exercises used in the resistance exercise 1)Standing chess press;(2)Strengthening back muscles in sitting position;(3)Standing strengthening abduction of both shoulders;(4)Standing strengthening flexion of both shoulders;(5)Standing strengthening flexion of both forearms;(6)Standing strengthening extension of both forearms;(7)Strengthening extension of both knees in sitting position;(8)Strengthening flexion of both knees in sitting position;(9)Strengthening dorsiflexion of both ankles in sitting position.
  Arms: Progressive resistance training
Other: Control group — The participants will receive information regarding health education.
  Arms: Control group

SUMMARY:
The study will be a randomized clinical trial and will be conducted in Civil Hospital and Kalsoom Hospital Samundry. This study will be completed in time duration of 10 months after the approval of synopsis. Non probability convenience sampling with Randomization technique will be used and 26 participants will be recruited in study after randomization. The subjects will be divided into two groups and the group A will receive Progressive training and Health education and group B will receive only Health education. The data will be assessed at the baseline and after 8th week of treatment. After data collection data will be analyzed by using SPSS version 21.

DETAILED DESCRIPTION:
The significance of this study is that it may improve the postmenopausal symptoms like depression and vasomotor symptoms which includes hot flushes , night sweats etc .in postmenopausal females. The majority of studies examining the vasomotor symptoms affected by symptoms of post menopause have concentrated on the effects of therapies like hormone therapy.To our knowledge, no studies have looked at the connection between vasomotor symptoms,depression and resistance training. Without doing so, it is challenging to understand how Vasomotor symptoms have an impact. This study sought to fill in the knowledge vaccum by examining the resistance training effect on depression , fatigue and vasomotor symptoms.

ELIGIBILITY:
Inclusion Criteria:

Post-menopausal women with age 50 - 60 years Blood pressure less than 160 / 100 More than or equal to 4 moderate-severe vasomotor symptoms including hot flushes, nocturnal sweats, sweating and poor sleep.

Exclusion Criteria:

Chronic metabolic and endocrine diseases Receiving hormone replacement treatment Surgical menopause Cognitive impairment

Ages: 50 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 64 (Estimated)
Dates: Start 2023-04-05 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-10 (Estimated)

PRIMARY OUTCOMES:
Hot Flash related Interference Scale (HFRDIS) for vasomotor symptoms | 6th week
  The HFRDIS is a 10-item scale which measures the degree hot flashes interfere with daily activities; the tenth item measures the degree hot flashes interfere with overall quality of life. The HFRDIS was internally consistent, with alphas of 0.96 at times
FATIGUE SEVERITY SCALE | 6th week
  The Fatigue Severity Scale (FSS) is a 9-item scale which measures the severity of fatigue and its effect on a person's activities and lifestyle.
DASS-21( Depression, Anxiety and stress scale 21-item | 6th Week
  DASS-21 is a self reported questionnaire which is used to assess the severity of range of symptoms like depression, anxiety and stress. It is not only used to measure the severity of symptoms but can also be used to assess the subject's response to treatment.The reliability of DASS-21 showed that it has excellent Cronbach's alpha values of 0.81,0.89 and 0.78 for the subscales of depressive, anxiety and stress respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- Civil Hospital Samundry, Samundry, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Daley A, Stokes-Lampard H, Thomas A, MacArthur C. Exercise for vasomotor menopausal symptoms. Cochrane Database Syst Rev. 2014 Nov 28;2014(11):CD006108. doi: 10.1002/14651858.CD006108.pub4. PMID 25431132
- [Background] Ivarsson T, Spetz AC, Hammar M. Physical exercise and vasomotor symptoms in postmenopausal women. Maturitas. 1998 Jun 3;29(2):139-46. doi: 10.1016/s0378-5122(98)00004-8. PMID 9651903
- [Background] Berin E, Hammar M, Lindblom H, Lindh-Astrand L, Spetz Holm AC. Effects of resistance training on quality of life in postmenopausal women with vasomotor symptoms. Climacteric. 2022 Jun;25(3):264-270. doi: 10.1080/13697137.2021.1941849. Epub 2021 Jul 9. PMID 34240669